CLINICAL TRIAL: NCT05543460
Title: Assessment of Miniscrew-assisted Rapid Palatal Expansion With and Without Corticopuncture in Adults: A Randomized Clinical Trial
Brief Title: Miniscrew-assisted Rapid Palatal Expansion With and Without Corticopuncture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Yomna Mohamed Mohamed Yacout, Lecturer, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0489-8/2022
Record Dates: First submitted 2022-09-14; First posted 2022-09-16 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2022-09

CONDITIONS: Palatal Expansion Technique; Posterior Crossbite; Maxillary Hypoplasia; Malocclusion
Keywords: Rapid palatal expansion; Maxillary Skeletal Expander; Corticopunctures; MARPE
MeSH Terms: conditions — Retrognathia; Malocclusion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Corticopuncture-facilitated MARPE (Experimental): Patients will be treated using Maxillary Skeletal Expander (MSE II, Biomaterials Korea Inc., Seoul, Korea) with corticopunctures .along the mid-palatal suture
  Interventions: Procedure: MARPE with Corticopunctures
- Conventional MARPE (Active Comparator): Patients will be treated using Maxillary Skeletal Expander (MSE II, Biomaterials Korea Inc., Seoul, Korea) without corticopunctures.
  Interventions: Device: MARPE

INTERVENTIONS:
Procedure: MARPE with Corticopunctures — Maxillary Skeletal Expander (MSE II, Biomaterials Korea Inc., Seoul, Korea) used to correct the maxillary transverse deficiency aided with corticopunctures made along the mid-palatal suture
  Arms: Corticopuncture-facilitated MARPE
Device: MARPE — Maxillary Skeletal Expander (MSE II, Biomaterials Korea Inc., Seoul, Korea) used to correct the maxillary transverse deficiency
  Arms: Conventional MARPE

SUMMARY:
Rapid palatal expansion aims at skeletally correcting the transverse maxillary deficiency by applying forces to separate the mid-palatal suture. In adult patients, the separation of the mid-palatal suture may not be possible due to its increased interdigitation. Miniscrew-assisted rapid maxillary expansion (MARPE) was proposed to transmit the forces directly to the mid-palatal suture through palatal miniscrews in addition to the anchor teeth. However, some non-growing patients may not respond favorably to MARPE. Hence, the use of corticopunctures as an adjunct to MARPE was recently proposed to overcome the increased resistance of the sutures in adult patients.

The study aims to assess and compare the skeletal and dental effects of miniscrew-assisted rapid palatal expansion with and without corticopunctures in non-growing patients.

DETAILED DESCRIPTION:
Rapid palatal expansion is a common treatment modality that aims at skeletally correcting the transverse maxillary deficiency by applying forces to separate the mid-palatal suture. In adult patients, the separation of the mid-palatal suture may not be possible due to its increased interdigitation and ossification. Miniscrew-assisted rapid maxillary expansion (MARPE) was proposed to transmit the forces directly to the mid-palatal suture through palatal miniscrews in addition to the anchor teeth. However, some non-growing patients may not respond favorably to MARPE. Hence, the use of corticopunctures as an adjunct to MARPE was recently proposed to overcome the increased resistance of the ossified mid-palatal sutures in adult patients.

The aim of the study is to assess and compare the skeletal and dental effects of miniscrew-assisted rapid palatal expansion with and without corticopunctures in non-growing patients.

A randomized clinical trial will be conducted to address the aim of the study. Patients will be randomly and equally assigned to group 1 (Corticopuncture-facilitated MARPE) or group 2 (Conventional MARPE). Both groups will be treated using Maxillary Skeletal Expander (MSE II, Biomaterials Korea Inc., Seoul, Korea). Ten corticopunctures will be made in group 1 along the mid-palatal suture with the aid of a 3D printed surgical guide. The skeletal and dental changes will be assessed using cone beam computed tomography scans obtained before treatment and after 6 months of expansion stabilization. The results will be compared between the groups and analyzed using the appropriate statistical tests.

ELIGIBILITY:
Inclusion Criteria:

1. Suture maturation stage D or E according to the method of Angelieri et al. (Angelieri F, Cevidanes LH, Franchi L, Goncalves JR, Benavides E, McNamara JA, Jr. Midpalatal suture maturation: classification method for individual assessment before rapid maxillary expansion. Am J Orthod Dentofacial Orthop. 2013;144(5):759-69.)
2. Maxillary transverse deficiency measured using the method of Cantarella et al. (Cantarella D, Dominguez-Mompell R, Mallya SM, Moschik C, Pan HC, Miller J, et al. Changes in the midpalatal and pterygopalatine sutures induced by micro-implant-supported skeletal expander, analyzed with a novel 3D method based on CBCT imaging. Prog Orthod. 2017;18(1):34.)
3. Good oral hygiene (Score <2 based on the Simplified Oral Hygiene Index (OHI-S)). (Greene JC, Vermillion JR. The Simplified Oral Hygiene Index. J Am Dent Assoc. 1964;68:7-13.)

Exclusion Criteria:

1. History of previous orthodontic or orthopedic treatment.
2. History of facial trauma or surgery.
3. Patients with congenital craniofacial malformations or diagnosed syndromes.
4. Medical history that prohibits the surgical intervention.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Transverse skeletal changes from baseline to an average of 6 months after the initial activation, measured using cone beam computed tomography (CBCT) | At baseline and an average of 6 months after the initial activation
  The data from CBCT scans at the different time points will be exported in Digital Imaging and Communications in Medicine (DICOM) format and processed using suitable software. The relevant landmarks will be defined and located by the investigator to measure the transverse skeletal changes in mm from baseline to the end of passive retention of the expansion.

SECONDARY OUTCOMES:
Dento-alveolar inclination changes from baseline to an average of 6 months after the initial activation, measured using CBCT | At baseline and an average of 6 months after the initial activation
  The data from CBCT scans at the different time points will be exported in DICOM format and processed using suitable software. The relevant landmarks will be defined and located by the investigator to measure the changes in dentoalveolar inclination from baseline to the end of passive retention of the expansion.

CONTACTS AND LOCATIONS:
Overall Officials: Yomna M Yacout, MSc, PhD, Principal Investigator — Alexandria University; Eiman S Marzouk, MSc, PhD, Study Chair — Alexandria University
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zeuke W, Heidrich R. [Late paralysis of the peripheral nerves from the neurologic viewpoint]. Zentralbl Neurochir. 1983;44(1):53-5. German. PMID 6305058
- [Background] Bud ES, Bica CI, Pacurar M, Vaida P, Vlasa A, Martha K, Bud A. Observational Study Regarding Possible Side Effects of Miniscrew-Assisted Rapid Palatal Expander (MARPE) with or without the Use of Corticopuncture Therapy. Biology (Basel). 2021 Mar 3;10(3):187. doi: 10.3390/biology10030187. PMID 33802266
- [Background] Angelieri F, Cevidanes LH, Franchi L, Goncalves JR, Benavides E, McNamara JA Jr. Midpalatal suture maturation: classification method for individual assessment before rapid maxillary expansion. Am J Orthod Dentofacial Orthop. 2013 Nov;144(5):759-69. doi: 10.1016/j.ajodo.2013.04.022. PMID 24182592
- [Background] Cantarella D, Dominguez-Mompell R, Mallya SM, Moschik C, Pan HC, Miller J, Moon W. Changes in the midpalatal and pterygopalatine sutures induced by micro-implant-supported skeletal expander, analyzed with a novel 3D method based on CBCT imaging. Prog Orthod. 2017 Nov 1;18(1):34. doi: 10.1186/s40510-017-0188-7. PMID 29090368
- [Background] GREENE JC, VERMILLION JR. THE SIMPLIFIED ORAL HYGIENE INDEX. J Am Dent Assoc. 1964 Jan;68:7-13. doi: 10.14219/jada.archive.1964.0034. No abstract available. PMID 14076341